CLINICAL TRIAL: NCT01595321
Title: Pilot Study Evaluating Allogeneic GM-CSF-Transduced Pancreatic Tumor Cell Vaccine (GVAX) and Low Dose Cyclophosphamide With Fractionated Stereotactic Body Radiation Therapy (SBRT) and FOLFIRINOX Chemotherapy in Patients With Resected Adenocarcinoma of the Pancreas
Brief Title: Pancreatic Tumor Cell Vaccine (GVAX), Cyclophosphamide, SBRT, and FOLFIRINOX in Patients With Resected Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: The Skip Viragh Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J1179; NA_00050233 (Other: JHMIRB)
Record Dates: First submitted 2012-04-27; First posted 2012-05-10 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer
Keywords: Adjuvant therapy; Immunotherapy; Cytoxan; Cyclophosphamide; Pancreatic Vaccine; Stereotactic radiation therapy; SBRT; FOLFIRINOX; GVAX
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; Radiosurgery; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1: SBRT and FOLFIRINOX (Experimental): The initial 3 patients were treated with SBRT and full dose FOLFIRINOX and observed for the first 2 cycles (8 weeks) for dose limiting toxicities (DLTs). If 2-3 patients are observed with uncontrolled grade 3-4 diarrhea, 2-3 patients are observed with grade 3-4 thrombocytopenia, or if 3 patients are observed with grade 3-4 neutropenia within the first 2 cycles of FOLFIRINOX administration (8 weeks) then the dose level will be deemed unacceptable.
  Interventions: Radiation: Stereotactic Body Radiation; Drug: FOLFIRINOX
- Cohort 2: SBRT and modified FOLFIRINOX (Experimental): The next 4 patients were treated with SBRT and modified FOLFIRINOX and observed for the first 2 cycles (8 weeks) for dose limiting toxicities (DLTs). If no patients are observed with grade 3-4 diarrhea, thrombocytopenia, or neutropenia, then the next cohort of patients will receive SBRT, modified FOLFIRINOX, and GVAX (with Cy).
  Interventions: Radiation: Stereotactic Body Radiation; Drug: FOLFIRINOX
- Cohort 3: CY, GVAX, SBRT, and modified FOLFIRINOX (Experimental): The last 12 patients will receive Cy, GVAX, SBRT, and modified FOLFIRINOX.
  Interventions: Drug: Cyclophosphamide; Biological: GVAX Pancreas Vaccine; Radiation: Stereotactic Body Radiation; Drug: FOLFIRINOX

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (Cy) 200 mg/m^2 administered one day prior to GVAX (day 0). One dose will be given prior to SBRT and FOLFIRINOX and four additional doses after FOLFIRINOX completion for a total of 5 doses. Additional CY/GVAX boosts may be given every 6 months thereafter until disease recurrence.
  Other Names: Cytoxan; Cy
  Arms: Cohort 3: CY, GVAX, SBRT, and modified FOLFIRINOX
Biological: GVAX Pancreas Vaccine — GVAX administered one day after Cy (day 1). One dose will be given prior to SBRT and FOLFIRINOX and four additional doses after FOLFIRINOX completion for a total of 5 doses. Additional CY/GVAX boosts may be given every 6 months thereafter until disease recurrence.
  Other Names: GVAX; PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1/GM-Neo vaccine
  Arms: Cohort 3: CY, GVAX, SBRT, and modified FOLFIRINOX
Radiation: Stereotactic Body Radiation — Cohort 1 and 2: SBRT (6.6 Gy per day, 33 Gy total dose) will be administered over 5 days within 6-10 weeks of pancreas surgery (Whipple).
  Cohort 3: SBRT (6.6 Gy) will be administered over 5 days starting between 13-17 days after the first dose of CY/GVAX.
  Other Names: SBRT
Drug: FOLFIRINOX — FOLFIRINOX is given over six 28-day cycles, starting at least 1 weeks after SBRT.
  FOLFIRINOX consists of the following drugs given IV on days 1 and 15 of each cycle:
  Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (400 mg/m^2 bolus followed by 2,400 mg/m^2 continuous infusion over 46-48 hours);
  modified FOLFIRINOX consists of the same regimen described above but without the 400 mg/m^2 Fluorouracil bolus.

SUMMARY:
The purpose of this study is to estimate safety of GVAX Pancreas Vaccine (GVAX) with immune modulating doses of cyclophosphamide (Cy) followed by SBRT and FOLFIRINOX chemotherapy in pancreatic cancer patients after surgery.

DETAILED DESCRIPTION:
This study enrolled patients with surgically resected adenocarcinoma of the pancreas who had titanium clips placed at the time of surgery in order to guide SBRT treatment.

Enrollment was based on traditional 3+3 design with grade 3-4 diarrhea and/or neutropenia defined as the dose limiting toxicity (DLT) within the first 2 cycles (8 weeks) of FOLFIRINOX. The first group of 3 patients (Cohort 1) received SBRT and full dose FOLFIRINOX. The second group of 4 patients (Cohort 2) received SBRT and modified FOLFIRINOX, and the third group of 12 patients (Cohort 3) received SBRT and modified FOLFIRINOX as well as Cy/GVAX vaccinations.

Cy/GVAX (patients 8-19): cyclophosphamide (Cy) at 200 mg/m^2 intravenously over 30 minutes the day before each vaccine. Each vaccination (GVAX) consists of six total intradermal injections of vaccine, two each in the upper right and left thighs, and two in the upper non-dominant arm. Each injection consists of approximately 2.5x10^8 cells of each cell line (PANC 6.03/PANC 10.05) for a total of 5x10^8 cells. The first dose of Cy/GVAX was given within 6-10 weeks from surgery.

Adjuvant SBRT was given 13-17 days after the first dose of Cy/GVAX. Patients receive 5 days of SBRT (6.6 gray (Gy) daily for 33 Gy total) to the tumor bed as delineated by surgical clips placed by the surgeon.

Six 28-day cycles of FOLFIRINOX, starting at least one week after completion of SBRT.

This was permitted to be given locally. Patients were evaluated for dose limiting toxicities (DLTs) within the first 2 cycles (8 weeks).

Cy/GVAX #2-5 was given every 28 days (+/- 3 days), starting 35 days (+/- 7 days) after completion of FOLFIRINOX. Patients without evidence of recurrence could then qualify for additional Cy/GVAX boosts every 6 months (every 12 months with Amendment #10) until disease recurrence, toxicity, withdrawal, or death.

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Documented cancer of the pancreas (head, neck, and/or uncinate process), that has been completely resected
2. No prior Chemotherapy, radiation therapy or biologic therapy for pancreatic cancer
3. Must be within 10 weeks from surgical resection of cancer
4. Titanium clips (minimum 1) must be placed at the time of surgery to aid in SBRT treatment planning
5. ECOG Performance Status of 0 to 1
6. Adequate organ function as defined by study-specified laboratory tests
7. Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
8. Signed informed consent form
9. Willing and able to comply with study procedures

Exclusion criteria (abbreviated):

1. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
2. Presence of metastatic disease
3. Clinical metabolic or laboratory abnormalities defined as Grade 3 or 4 of the National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0
4. Systemically active steroids
5. Chemotherapy, radiation therapy or biologic therapy within 28 days prior to receiving study drug
6. Inability to begin protocol treatment within 70 days (10 weeks) after surgery to remove cancer
7. History of HIV, hepatitis B or C infection
8. Pregnant or lactating
9. Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laheru, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: SBRT and FOLFIRINOX: Stereotactic Body Radiation Therapy (SBRT, 33 Gy cumulative dose) was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of FOLFIRINOX were given starting 7-28 days after completion of SBRT. Full dose FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle): Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (400 mg/m^2 bolus followed by 2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions of FOLFIRINOX were permitted.
- Cohort 2: SBRT and Modified FOLFIRINOX: Stereotactic Body Radiation Therapy (SBRT), 33 Gy cumulative dose, was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of modified FOLFIRINOX were given, starting 7-28 days after completion of SBRT. Modified FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle): Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions were permitted.
  The difference between Cohort 1 and 2 is that the Fluorouracil bolus was dropped in Cohort 2.
- Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX: Cyclophosphamide: Cyclophosphamide (CY) 200 mg/m^2 was administered one day prior to GVAX (day 0). GVAX Pancreas Vaccine (GVAX) will be administered one day after CY (day 1). One Cycle of Cy/GVAX was given prior to SBRT and FOLFIRINOX and four additional doses after FOLFIRINOX completion for a total of 5 doses. Additional CY/GVAX boosts were given every 6 months thereafter until disease recurrence.
  Stereotactic Body Radiation Therapy (SBRT), 33 Gy cumulative dose, was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of modified FOLFIRINOX were given, starting 7-28 days after completion of SBRT. Modified FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle): Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions were permitted.
Period: Overall Study
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Started | 3 | 4 | 12
Completed (Completed = received all planned doses of SBRT + FOLFIRINOX (Cohorts 1 and 2), or all planned doses of SBRT + FOLFIRINOX and all 5 monthly cycles of Cy and GVAX (Cohort 3)) | 2 | 3 | 7
Not Completed | 1 | 1 | 5
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: SBRT and FOLFIRINOX: Stereotactic Body Radiation Therapy (SBRT, 33 Gy cumulative dose) was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of FOLFIRINOX were given starting 7-28 days after completion of SBRT. Full dose FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (400 mg/m^2 bolus followed by 2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions of FOLFIRINOX were permitted.
- Cohort 2: SBRT and Modified FOLFIRINOX: Stereotactic Body Radiation Therapy (SBRT, 33 Gy cumulative dose) was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of modified FOLFIRINOX were given, starting 7-28 days after completion of SBRT. Modified FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions of FOLFIRINOX were permitted.
  The difference between Cohort 1 and 2 is that the Fluorouracil bolus was dropped in Cohort 2.
- Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX: Cyclophosphamide (Cy) 200 mg/m^2 was administered on Day 0 of each vaccine cycle. GVAX Pancreas Vaccine (GVAX) was administered one day after Cy (Day 1 of each cycle). The first Cycle of Cy/GVAX was given 6-10 weeks after pancreas surgical resection (prior to SBRT and FOLFIRINOX). Four additional doses were given after FOLFIRINOX completion for a total of 5 priming doses. Additional Cy/GVAX boosts were given every 6 months thereafter until disease recurrence.
  Stereotactic Body Radiation Therapy (SBRT), 33 Gy cumulative dose, was administered to the surgical bed over 5 days, starting about 2 weeks after the first dose of Cy/GVAX.
  Six 28-day cycles of modified FOLFIRINOX were given, starting 7-28 days after completion of SBRT. Modified FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions were permitted.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX | Total
Number analyzed (Participants) | 3 | 4 | 12 | 19
Age, Continuous [Median (Full Range); unit: years] | 69 [63 to 73] | 55 [50 to 65] | 58 [41 to 69] | 58 [41 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 6
  Male | 3 | 2 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 12 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 4 | 12 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Classification [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5: 0= fully active, performs without restrictions, 1= can ambulate, but restricted in physical strenuous activity, 2= ambulatory and capable of self-care but unable to work, active for >50%of waking hours, 3= limited self-care, confined to bed or chair for >50%of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    ECOG 0 | 2 | 2 | 7 | 11
    ECOG 1 | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: The number of participants experiencing grade 3-4 diarrhea, neutropenia, and thrombocytopenia within the first 2 cycles (8 weeks) of treatment, regardless of attribution. The rates of each of these toxicities were considered unacceptable if they were 40%, 60%, and 40%, respectively. A decision rule similar to the traditional 3+3 design was used to determine whether it was safe to continue on to the next cohort.
Time Frame: 8 weeks
Population: One patient in cohort 2 was not evaluable because they did not complete 2 cycles of FOLFIRINOX.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: SBRT and Modified FOLFIRINOX: Stereotactic Body Radiation Therapy (SBRT), 33 Gy cumulative dose, was administered to the surgical bed over 5 days, starting 6-10 weeks after pancreas surgical resection (Whipple procedure).
  Six 28-day cycles of modified FOLFIRINOX were given, starting 7-28 days after completion of SBRT. Modified FOLFIRINOX consists of the following drugs, given IV on Days 1 and 15 of each cycle: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). Dose reductions were permitted.
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 3 | 3 | 12
Participants
  Diarrhea | 0 | 0 | 1
  Neutropenia | 3 | 0 | 1
  Thrombocytopenia | 2 | 0 | 0

2. Primary Outcome: Grade 3 or Higher Cy/GVAX-related Adverse Events
Description: Number of participants with grade 3 or above adverse event attributed to Cy or the GVAX pancreas vaccine. Each adverse event (as defined by NCI CTCAE v4.0) was counted only once for a given subject.
Time Frame: 116 months
Population: Only Cohort 3 received Cy and GVAX and could be evaluated for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 12
Participants | 2

3. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the amount of time from date of surgery until death or end of follow-up. OS was censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 96 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 3 | 4 | 12
months | 22.2 [6.74 to NA] — upper limit goes to infinity | 27.5 [16.3 to NA] — upper limit goes to infinity | 61.3 [11.1 to NA] — upper limit goes to infinity

4. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS was measured as the time from date of surgery until pancreatic cancer recurrence or death. Disease status was monitored by radiologic scans done approximately every 12 weeks. DFS was censored on the date of last radiologic scan for subjects without documentation of cancer recurrence or death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 96 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 3 | 4 | 12
months | 10.5 [3.45 to NA] — upper limit goes to infinity | 14.5 [10.1 to NA] — upper limit goes to infinity | 24.1 [11.1 to NA] — upper limit goes to infinity

5. Secondary Outcome: Distant Metastases Free Survival (DMFS)
Description: DMFS was measured as the amount of time from date of surgery until metastatic disease progression or death. Metastatic disease progression is the appearance of one or more new lesions outside the primary tumor area (pancreas). Disease status was monitored by radiologic scans done approximately every 12 weeks. DMFS was censored on the date of last radiographic scans for subjects without documentation of metastatic disease progression or death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 96 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 3 | 4 | 12
months | 10.5 [3.45 to NA] — upper limit goes to infinity | 19.0 [10.15 to NA] — upper limit goes to infinity | 42.0 [11.1 to NA] — upper limit goes to infinity

6. Secondary Outcome: Freedom From Local Progression (FFLP)
Description: FFLP was measured as the time from date of surgery until disease recurrence in the pancreas or death. Disease status was monitored by radiologic scans done approximately every 12 weeks. FFLP was censored on the date of last radiographic scans for subjects without documentation of local disease recurrence or death at the time of analysis. Estimation based on the Kaplan-Meier curve.
Time Frame: 96 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
Number analyzed (Participants) | 3 | 4 | 12
months | 17.3 [6.74 to NA] — upper limit goes to infinity | 20.5 [10.8 to NA] — upper limit goes to infinity | 34.0 [11.1 to NA] — upper limit goes to infinity

ADVERSE EVENTS:
Time Frame: 116 months
Groups:
- Cohort 1: SBRT and FOLFIRINOX: Stereotactic Body Radiation (SBRT, 6.6 Gy) will be administered over 5 days within 6-10 weeks of surgery (Whipple).
  FOLFIRINOX: FOLFIRINOX consist of the following: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (400 mg/m^2 bolus followed by 2,400 mg/m^2 continuous infusion over 46-48 hours). FOLFIRINOX will be administered over 6 cycles (Days 1 and 15 of each cycle) starting 7-28 days following completion of SBRT. Each cycle is 28 days long.
- Cohort 2: SBRT and Modified FOLFIRINOX: Stereotactic Body Radiation (SBRT, 6.6 Gy) will be administered over 5 days within 6-10 weeks of surgery (Whipple).
  FOLFIRINOX: FOLFIRINOX consist of the following: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). FOLFIRINOX will be administered over 6 cycles (Days 1 and 15 of each cycle) starting 7-28 days following completion of SBRT. Each cycle is 28 days long.
  The difference between Cohort 1 and 2 is that the Fluorouracil bolus was dropped in Cohort 2.
- Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX: Cyclophosphamide: Cyclophosphamide (CY) 200 mg/m^2 will be administered one day prior to GVAX (day 0). One dose will be given prior to SBRT and FOLFIRINOX and four additional doses after FOLFIRINOX completion for a total of 5 doses. Additional CY/GVAX boosts may be given every 6 months thereafter until disease recurrence.
  GVAX Pancreas Vaccine: GVAX will be administered one day after CY (day 1). One dose will be given prior to SBRT and FOLFIRINOX and four additional doses after FOLFIRINOX completion for a total of 5 doses. Additional CY/GVAX boosts may be given every 6 months thereafter until disease recurrence.
  Stereotactic Body Radiation (SBRT, 6.6 Gy) will be administered over 5 days starting between 13-17 days after the first dose of CY/GVAX.
  FOLFIRINOX: FOLFIRINOX consist of the following: Oxaliplatin (85 mg/m^2), Irinotecan (180 mg/m^2), Leucovorin (400 mg/m^2), Fluorouracil (2,400 mg/m^2 continuous infusion over 46-48 hours). FOLFIRINOX will be administered over 6 cycles (Days 1 and 15 of each cycle) starting 7-28 days following completion of SBRT and at least 28 days after the first vaccine. Each cycle is 28 days long.
Arm/Group | Cohort 1: SBRT and FOLFIRINOX | Cohort 2: SBRT and Modified FOLFIRINOX | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/4 | 8/12
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/4 | 6/12
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SBRT and FOLFIRINOX (N=3) | Cohort 2: SBRT and Modified FOLFIRINOX (N=4) | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter realted infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction, partial (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: SBRT and FOLFIRINOX (N=3) | Cohort 2: SBRT and Modified FOLFIRINOX (N=4) | Cohort 3: CY, GVAX, SBRT, and Modified FOLFIRINOX (N=12)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (5) | 8 (9)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 1 (2) | 1 (1)
Annuloaortic ectasia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 6 (8)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5)
Arthritis (gout) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ascities (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Blood and lymphativ system disorders, lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Bruising (vaccine site) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 3 (3) | 1 (2) | 5 (8)
Cold intolerance (General disorders) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (3) | 3 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Coronary arterial calcification (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (15) | 3 (7) | 10 (24)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 7 (7)
Dry Lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 6 (11)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 5 (5)
Erythema mutliforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Eye disorder (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (4) | 3 (6) | 11 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (2) | 1 (2) | 6 (11)
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (5)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 4 (7)
Gall bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gall bladder obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrointestinal disorders- others, specify (dark stools) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (6) | 4 (5)
Hearing imaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hematoma, liver (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma, Mediport (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 6 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 2 (2) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 3 (5) | 5 (6)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5) | 1 (4) | 6 (21)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Mucoasal infection (Infections and infestations) | 0 (0) | 1 (2) | 3 (3)
Mucositis (oral ulcers) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (6) | 8 (15)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0) | 3 (6)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (3) | 2 (4) | 7 (9)
Pallor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 4 (5) | 10 (11)
Photophobia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (5) | 1 (2) | 4 (13)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pneumobilia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 5 (10)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (4)
Renal cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder - other, tracheal deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 3 (3)
Skin and Subcutaneous Tissue disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 6 (6)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin tears (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction, partial (Gastrointestinal disorders) | 1 (1) | 1 (5) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thymic hyperplasia (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vertebral compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Ventricular gallop (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2) | 4 (6)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (4) | 0 (0) | 6 (11)
White blood (Investigations) | 2 (2) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3)
Erythema (Vaccine site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 12 (63)
Induration (Vaccine Site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 12 (65)
Prutitus (Vaccine site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (54)
Skin discoloration (Vaccine Site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (6)
Tenderness (Vaccine Site) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 9 (26)
Vaccine Site Flares (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (11)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT01595321/Prot_SAP_000.pdf